CLINICAL TRIAL: NCT05532527
Title: Efficacy and Safety of Microwave Ablation Combined With Camrelizumab and Chemotherapy in Patients With Advanced Non-small Cell Lung Cancer: a Multicenter, Open, Prospective Study
Acronym: NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-MWA-001
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Microwave ablation combined with Camrelizumab and chemotherapy
  Interventions: Drug: Microwave ablation combined with Camrelizumab and chemotherapy

INTERVENTIONS:
Drug: Microwave ablation combined with Camrelizumab and chemotherapy — Microwave ablation combined with Camrelizumab and chemotherapy
  Other Names: Camrelizumab

SUMMARY:
To evaluate the efficacy and safety of microwave ablation combined with Camrelizumab and chemotherapy in the treatment of patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1.Have fully understood and voluntarily signed the informed consent for this study 2.18-75 years old 3.Stage IIIB-IV non-small cell lung cancer patients with histologically or cytologically confirmed EGFR/ALK- 4.No previous systemic antitumor therapy for the target lesion 5.ECOG score is 0-2 6.The predicted survival time was ≥3 months 7.At least one measurable lesion (according to RECIST 1.1) other than the lesion that underwent microwave ablation 8.The function of major organs is normal, and the test results during screening must meet the following requirements:

1. Blood routine (no blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte macrophage colony-stimulating factor (GM-CSF) treatment within 14 days before screening) :

   A. Hemoglobin (Hb) ≥ 90 g/L; B. Neutrophil count (ANC) ≥ 1.5×109/L; C. Platelet count (PLT) ≥ 80 ×109/L;
2. Biochemical tests shall meet the following standards:

   A. Total bilirubin (TBIL) < 1.5 ULN; B. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 ULN and < 5 ULN in patients with liver metastases; C. Serum creatinine (Cr) ≤ 1.5 ULN or endogenous creatinine clearance > 50ml/min (cockcroft-gault formula); D. Urine routine test results showed urinary protein (UPRO) < 2+ or 24-hour urinary protein quantification <1g;
3. Echocardiography: left ventricular ejection fraction (LVEF) ≥50%;
4. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN; 9. Contraception: Women of reproductive age should agree that they must use effective contraception during and for 6 months after the study; Had a negative serum or urine pregnancy test within 7 days before study enrollment and had to be non-lactating; Men should agree to use contraception during the study and for 6 months after the end of the study

Exclusion Criteria:

1. Allergic to treatment drugs;
2. EGFR/ALK mutation positive;
3. There are high risk factors for local treatment complications such as bleeding, fistula and perforation;
4. Patients with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonitis and severe pulmonary function impairment (maximum volume < 40%);
5. Patients with coagulopathy who have severe bleeding tendency and cannot be corrected in a short time (prothrombin time >18 s, prothrombin activity <40%);
6. Anticoagulant therapy and/or antiplatelet drugs (except dabigatran, rivaroxaban and other new oral anticoagulants) were stopped for no more than 5 to 7 days before ablation.
7. Extensive pleural metastases with massive pleural effusion;
8. Patients with active brain metastases: untreated, newly diagnosed and/or growing lesions or symptomatic brain metastases (patients with stable symptoms after treatment of brain metastases were eligible to remain stable for at least 4 weeks);
9. Infection and radiation inflammation around the lesion, skin infection at the puncture site without good control, systemic infection, high fever >38.5 ℃;
10. Subjects with active autoimmune disease or a history of autoimmune disease, or active hepatitis B/C. Note: Subjects with hepatitis B who met the following criteria were also eligible for inclusion: The HBV viral load must be less than 104 copies per milliliter (2000IU per milliliter) before the first dose, and subjects should receive anti-hbv therapy to avoid virus reactivation throughout the study drug treatment. For subjects with anti-HBC (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required；
11. Patients were using immunosuppressive agents or systemic hormone therapy (dose >10mg/ day prednisone or other efficacy hormone) to achieve immunosuppression and continued to use them within 2 weeks before enrollment;
12. Has had or is currently suffering from other malignant tumours within 5 years, except cured cervical carcinoma in situ, non-melanoma skin cancer or other tumours/cancers that have undergone radical treatment and have shown no signs of disease for at least 5 years; 65/5000
13. Had received antitumor drug therapy (e.g., chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy, etc.) 4 weeks before or within 4 weeks of the first dose, with the exception of palliative radiotherapy to bone for pain relief;
14. Had undergone major surgery within 4 weeks before the first dose or was expected to undergo major surgery during the study;
15. Patients whose imaging showed that the tumor had invaded important blood vessels or who were judged by the investigator to be highly likely to invade important blood vessels during the subsequent study and cause fatal massive bleeding;
16. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months before enrollment; New York Heart Association (NYHA) grade of congestive heart failure ≥2; Arrhythmia (including QTc interval ≥ 450 ms in men and ≥ 470 ms in women); Left ventricular ejection fraction (LVEF) <50%;
17. Those who have a history of psychotropic drug abuse and are unable to quit or have mental disorders;
18. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
19. Those who received live attenuated vaccine within 30 days of the first dose or expected to receive live attenuated vaccine during the study period;
20. The subject has received or plans to receive solid organ or blood transplantation (except corneal transplantation) during the study;
21. Patients deemed ineligible for enrollment in the investigator's judgment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-09-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 24 months
  Progression free survival

SECONDARY OUTCOMES:
OS | Up to 24 months
  Overall survival
ORR | Up to 24 months
  Objective Response Rate
safety | Up to 24 months
  AE

OTHER OUTCOMES:
Immune function | Up to 24 months
  T lymphocyte

IPD SHARING:
Plan to Share IPD: No